CLINICAL TRIAL: NCT04794400
Title: The Application of a Mask in Patients With Severe Covid-19 Already Treated With High-flow Nasal Cannula.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Gustav Torisson, Principal Investigator, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-07078
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Critical care; Non-invasive ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): An additional oxygen mask was applied for 30 minutes, in patients with ongoing HFNC treatment.
  Interventions: Other: oxygen mask

INTERVENTIONS:
Other: oxygen mask — All patients fulfilling inclusion criteria would be offered to test the intervention as part of their care. The intervention consisted only of a standardised way to evaluate this new clinical routine.

SUMMARY:
Patients with severe hypoxemic respiratory failure due to Covid-19 are often treated with oxygen delivered through a high-flow nasal cannula (HFNC). This is according to guidelines. We have made the clinical observation that oxygenation sometimes improves when a mask (e.g. oxygen mask or inhalation mask) is applied on top of the HFNC. This has quickly become a clinical routine at intermediary care units at our hospital, where patients with HFNC are offered to test the intervention (mask + HFNC) as part of clinical routine.

This study aims to evaluate this new routine in a standardised way.

DETAILED DESCRIPTION:
Patients with severe covid-19, treated with HFNC, will be approached for consent. If inclusion critera and no exclusion criteria are fulfilled, baseline measurements will be taken without mask, including arterial blood gas analysis (ABG)

Then a simple oxygen mask will be applied covering nose and mouth, without providing supplemental oxygen. After 30 minutes with mask + HFNC, new measurements will be taken, including ABG.

After 30 minutes, the mask is removed and when steady state occurs, new measurements will be taken, without ABG. Then, the patients could continue using the mask as part of clinical routine

ELIGIBILITY:
Inclusion Criteria:

* Verified Covid19 infection
* treatment with HFNC
* Estimated P/F ratio of ≤ 13 KPa

Exclusion Criteria:

* language barrier
* unable to provide consent
* risk of deterioration due to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 30 minutes
  Change in SaO2 in % from ABG with mask vs without mask

SECONDARY OUTCOMES:
Carbon dioxide | 30 minutes
  Change in PaCO2 in KPa from ABG with mask vs without mask
SpO2 | 60 minutes
  Change in peripherally measured oxygen saturation before, with and after mask
Respiratory rate | 30 minutes
  Change in respiratory rate (breaths/min) with mask vs without mask

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Torisson, PhD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No